CLINICAL TRIAL: NCT01142492
Title: Postmarketing Surveillance Study on the Extent to Which Patient Compliance is Influenced by Use of a Variable Titration Regimen at the Start of Treatment of Relapsing Multiple Sclerosis With Interferon Beta 1a (Rebif®)
Brief Title: A Postmarketing Surveillance (PMS) Study to Evaluate the Extent to Which Patient Compliance is Influenced by Use of a Variable Titration Regimen at the Start of Treatment of Relapsing Multiple Sclerosis (MS) With Interferon Beta 1a (Rebif®)
Acronym: TOURIMS
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr. Norbert Zessack/Head of Medicine BU Neurology, Merck Serono GmbH Germany, an affiliate of MerckKGaA, Darmstadt, Germany
Other Study IDs: IMP28157
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Interferon beta; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

INTERVENTIONS:
Drug: Interferon beta-1a — Subjects first received Interferon beta-1a at a dose of 22 µg x3 over a period of 4 weeks. An attempt was then made to increase the dose of interferon beta-1a to 44 µg x3 as a self-administered subcutaneous (s.c.) injection. If intolerable interferon-specific side effects or problems of acceptance occured, the treatment with Rebif 22 µg three times weekly was continued.
  Other Names: Rebif

SUMMARY:
This was an open-label, multicentric, prospective, post-marketing surveillance (PMS) study on the extent to which subject compliance is influenced by use of a variable titration regimen at the start of treatment of relapsing MS with Rebif.

DETAILED DESCRIPTION:
Interferon beta has become the treatment of choice in relapsing MS. In previous clinical studies, the interferon-beta 1a (Rebif) used within the scope of this PMS study has demonstrated significant efficacy in all aspects of treatment - magnetic resonance imaging (MRI) data, relapse rate, and progression of disability. The PRISMS-4 study demonstrated that treatment with Rebif reduces the frequency and severity of clinical relapses over 4 years and slows the progression of disability.

In order to achieve good subject compliance, it is important that the subject be given a realistic picture of the expected result of treatment and of the demands that will be made in connection with the treatment. Interferon beta cannot cure MS, however treatment with Rebif can reduce the number and severity of relapses and delay the progression of disability.

Rebif therapy is a long-term therapy. For this reason, subject may not feel any positive effects immediately, but instead may notice the benefits of treatment only after a considerable period of time. The early period after the start of treatment is considered to be crucial in terms of whether the treatment will be accepted and tolerated by the subject or whether unplanned cessation of treatment will occur.

OBJECTIVES

The principal objective of this PMS study was to provide subjects with the greatest possible degree of safety and support by means of optimal management in the first few weeks after the start of treatment or after the change from a different treatment regimen. This objective was to be achieved by, among other things, a flexible dose escalation regimen that took into account individual subjects' acceptance. It is precisely during this critical early phase of treatment, marked as it is by uncertainty, change, and in some cases problems of tolerability, that poor subject compliance occurs, leading in some cases to treatment dropouts.

Another question addressed in the study was related to the small number of subjects who after this initial phase could not tolerate Rebif therapy at the high dosage (44 µg x3). In these cases there was the option of a temporary dose reduction to the lower dosage (22 µg x3). The objective of this dose reduction was to avoid an unnecessary change of treatment regimen and thereby to make an important contribution to improving compliance. In the present PMS study, particular attention was paid to the question of subject compliance at the start of Rebif therapy. This applied both to Rebif-naive subjects and to subjects who were being switched to Rebif after receiving other forms of MS therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically diagnosed multiple sclerosis (MS) and relapses

Exclusion Criteria:

* Subjects with secondary progressive MS (SPMS) without relapses, pregnant or breastfeeding subjects, and subjects with contra- indications.
* Subjects with systemic concomitant diseases (e.g. diabetes, heart disease, liver disease, or renal disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A group of subjects with MS who were at the start of treatment with Rebif or switched to Rebif from other forms of MS therapy.
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Subjects' compliance to treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Norbert Zessack, Study Director — Merck Serono GmbH, Germany